CLINICAL TRIAL: NCT02653391
Title: Part A: a Prospective, Randomized, Double-masked, Vehicle Controlled, Paired-eye Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability and Efficacy of Elamipretide Topical Ophthalmic Solution in Subjects With Fuchs' Corneal Endothelial Dystrophy (FCED) Presenting With Mild to Moderate Corneal Edema Part B: a Prospective, Randomized, Double-masked, Vehicle Controlled, Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of Elamipretide Topical Ophthalmic Solution in Subjects With FCED Presenting With Mild to Moderate Corneal Edema.
Brief Title: A Study Investigating the Safety, Tolerability, and Efficacy of Elamipretide Topical Ophthalmic Solution for the Treatment of Fuchs' Corneal Endothelial Dystrophy (FCED)
Acronym: SPIFD-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIFD-101
Record Dates: First submitted 2015-12-20; First posted 2016-01-12 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Fuchs' Corneal Endothelial Dystrophy (FCED)
Keywords: Fuchs' Corneal Endothelial Dystrophy; FCED; Ocuvia™; MTP-131
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — Ophthalmic Solutions; arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Elamipretide 1.0% Ophthalmic Solution Part A (Cohort 1) (Experimental): Part A Each subject will receive one drop of elamipretide 1.0% ophthalmic solution BID in the randomly selected study eye (Cohort 1).
  Interventions: Drug: Part A Elamipretide 1.0% Ophthalmic Solution
- Elamipretide 3.0% Ophthalmic Solution Part B (Cohort 2) (Experimental): Part B Each subject will receive one drop of elamipretide 3.0% ophthalmic solution BID in both the right and left study eyes (Cohort 2).
  Interventions: Drug: Part B Elamipretide 3.0% Ophthalmic Solution
- Placebo A (Placebo Comparator): Part A: Each subject will receive one drop of vehicle solution BID in the paired eye of the randomly selected study eye (Cohort 1).
  Interventions: Drug: Part A Placebo
- Part B Placebo (Placebo Comparator): Part B Each subject will receive one drop of vehicle solution BID in both the right and left study eyes (Cohort 2).
  Interventions: Drug: Part B Placebo

INTERVENTIONS:
Drug: Part A Elamipretide 1.0% Ophthalmic Solution — Part A Each subject will receive one drop of elamipretide 1.0% ophthalmic solution BID in the randomly selected study eye.
  Other Names: MTP-131, Bendavia
  Arms: Elamipretide 1.0% Ophthalmic Solution Part A (Cohort 1)
Drug: Part B Elamipretide 3.0% Ophthalmic Solution — Part B Each subject will receive one drop of elamipretide 3.0% ophthalmic solution BID in both eyes.
  Other Names: MTP-131, Bendavia
  Arms: Elamipretide 3.0% Ophthalmic Solution Part B (Cohort 2)
Drug: Part A Placebo — Part A Each subject will receive one drop of vehicle ophthalmic solution BID in the paired eye of the randomly selected study eye.
  Arms: Placebo A
Drug: Part B Placebo — Part B: Each subject will receive one drop of vehicle ophthalmic solution BID in both eyes.
  Arms: Part B Placebo

SUMMARY:
This is a Phase 1/2 prospective, randomized, double-masked, and vehicle-controlled trial in two parts to evaluate the safety, tolerability, and efficacy of elamipretide topical ophthalmic solution in patients with Fuchs' Corneal Endothelial Dystrophy (FCED) presenting with mild to moderate corneal edema.

DETAILED DESCRIPTION:
This is a Phase 1/2 trial in two parts. Part A is a prospective, randomized, double-masked, vehicle controlled, paired-eye study in approximately 16 subjects to evaluate safety, tolerability and efficacy of elamipretide 1.0% topical ophthalmic solution in patients with Fuchs' Corneal Endothelial Dystrophy (FCED) presenting with mild to moderate corneal edema. Part B is a prospective, randomized double-masked, vehicle controlled study in approximately 11 subjects to evaluate safety, tolerability, and efficacy of elamipretide 3.0% topical ophthalmic solution in patients with FCED presenting with mild to moderate corneal edema.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old at the time of Screening Visit
* Diagnosis of FCED OU (both eyes) based on clinical and ophthalmic test findings
* Clinical evidence of corneal edema OU diagnosed with FCED, including one or more of the following signs: corneal epithelial microcysts, corneal epithelial bullae, stromal folds, or stromal haze
* Central corneal thickness of 550 μm to 700 μm (inclusive) in at least one eye diagnosed with FCED, as measured by ultrasonic pachymetry at the time of Screening Visit and Baseline Visit
* Best-corrected distance visual acuity (BCVA) of 20/25 to 20/320 (inclusive) at the time of Screening Visit and Baseline Visit OU
* Women of childbearing potential must agree to use birth control as specified in the protocol from the date they sign the informed consent form (ICF) until after the last study
* Able to give informed consent and willing to comply with all study visits and examinations
* Part B only: The presence of central endothelium, as determined by the investigator, with an area of contiguous endothelial cells within 1 mm of the central cornea as measured by confocal laser scanning microscopy (CLSM) or specular microscopy at the time of Screening Visit

Exclusion Criteria:

* Corneal findings of any type (including, but not limited to, stromal haze or stromal scarring), in either eye, that, based on investigator's assessment, limit the probability of visual improvement after corneal deturgescence
* Any ocular pathology requiring treatment with topical ophthalmic drops, with the exception of glaucoma or ocular hypertension
* Use of topical hypertonic saline drops for 3 days prior to Screening and throughout the duration of the study
* History of corneal disease (other than FCED) or corneal surgery in either eye
* Current use or likely need for the use of contact lens at any time during the study
* History of previous corneal or anterior segment surgery such as LASIK, photorefractive keratectomy, endothelial keratoplasty, penetrating keratoplasty cataract surgery or glaucoma surgery.
* Any disease or medical condition that in the opinion of the investigator would prevent the subject from participating in the study or might confound study results
* Participation in other investigational drug or device clinical trials within 30 days prior to enrollment, or planning to participate in any other investigational drug or device clinical trials within 30 days of study completion
* Women who are pregnant or lactating
* Part B only: Participation in Part A of SPIFD-101

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Raizman, MD, Principal Investigator — Ophthalmic Consultants of Boston; Edward Holland, MD, Principal Investigator — Cincinnati Eye Institute
Locations (2):
- United States (2):
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Ophthalmic Consultants of Boston, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A 18 participants were randomized. The treatment eye was chosen at random and the fellow eye was the control/placebo eye.
  Part B The participants received either treatment in both eyes or placebo in both eyes.
Units Other Than Participants: eyes
Groups:
- Elamipretide 1.0% Ophthalmic Solution and Placebo Part A (Cohort 1): Part A: Each subject will receive one drop of elamipretide 1.0% ophthalmic solution twice daily (BID) in the randomly selected study eye, and Placebo twice daily (BID) in the paired eye.
- Elamipretide 3.0% Ophthalmic Solution Part B (Cohort 2): Part B Each subject will receive one drop of elamipretide 3.0% ophthalmic solution twice daily (BID) in both the right and left study eyes (Cohort 2).
  Part B Elamipretide 3.0% Ophthalmic Solution
- Placebo Part B (Cohort 2): Part B Each subject will receive one drop of placebo comparator solution twice daily (BID) in both the right and left study eyes (Cohort 2).
  Placebo Part B
Period: Overall Study
Arm/Group | Elamipretide 1.0% Ophthalmic Solution and Placebo Part A (Cohort 1) | Elamipretide 3.0% Ophthalmic Solution Part B (Cohort 2) | Placebo Part B (Cohort 2)
Started | 18; 36 eyes | 3; 6 eyes | 1; 2 eyes
Completed | 16; 32 eyes | 1; 2 eyes | 1; 2 eyes
Not Completed | 2; 4 eyes | 2; 4 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Groups:
- Elamipretide 1.0% Ophthalmic Solution and Placebo: Part A participants includes those receiving Elamipretide and placebo
- Part B Elamipretide 3.0% Ophthalmic Solution: Part B Participants includes those receiving Elamipretide.
- Part B Placebo: Part B Participants include those receiving Placebo.
- Total: Total of all reporting groups
Arm/Group | Elamipretide 1.0% Ophthalmic Solution and Placebo | Part B Elamipretide 3.0% Ophthalmic Solution | Part B Placebo | Total
Number analyzed (Participants) | 18 | 3 | 1 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] — For Part B mean and Standard deviation data is not available; only range. Participants for Part B ranged between 58 and 70 years of age.
  years | 67.9 (8.64) | NA (NA) — For Part B, no summary statistics were calculated; mean and Standard deviation data is not available; only range. Participants for Part B ranged between 58 and 70 years of age. | NA (NA) — For Part B, no summary statistics were calculated; mean mean and Standard deviation data is not available; only range. Participants for Part B ranged between 58 and 70 years of age. | 67.9 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 1 | 10
  Male | 10 | 2 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 3 | 1 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 16 | 3 | 1 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Smoking [Count of Participants; unit: Participants] — Number of participants who formerly smoked
  Participants
    Former Smoker | 10 | 3 | 0 | 13
    Current Smoker | 1 | 0 | 0 | 1
    Never Smoker | 7 | 0 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular TEAEs.
Description: The incidence and severity of ocular treatment emergent adverse events (TEAEs)
Time Frame: Screening Visit, Baseline (Day 1), Week 1, Week 4, Week 8, Week 12, and Week 16
Population: All participants for whom ocular TEAEs were measured.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Placebo: Part A participants includes those receiving vehicle in eye paired with treatment eye.
- Part A Elamipretide 1.0% Ophthalmic Solution: Part A participants includes those receiving 1% Elamipretide
- Part B Placebo: Part B participants includes those receiving vehicle in both eyes.
- Part B Elamipretide 3.0% Ophthalmic Solution: Part B Participants includes those receiving 3% Elamipretide
Arm/Group | Part A Placebo | Part A Elamipretide 1.0% Ophthalmic Solution | Part B Placebo | Part B Elamipretide 3.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18 | 1 | 3
Participants
  Ocular mild TEAEs | 3 | 6 | 1 | 1
  Ocular moderate TEAEs | 0 | 0 | 0 | 2
  Ocular severe TEAEs | 0 | 0 | 0 | 0

2. Primary Outcome: The Incidence and Severity of Systemic Adverse Events
Description: The incidence and severity of systemic treatment emergent adverse events (TEAEs)
Time Frame: Screening Visit, Baseline (Day 1), Week 1, Week 4, Week 8, Week 12, and Week 16
Population: All participants for whom systemic TEAEs were measured. For Part A systemic events were not necessarily attributed to either intervention or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Elamipretide 1.0% Ophthalmic Solution or Placebo: Part A participants includes those receiving 1% Elamipretide in one eye and Placebo in paired eye.
- Part B Placebo: Part B Placebo includes participants who received vehicle only in both eyes.
- Part B Elamipretide 3.0% Ophthalmic Solution: Part B Participants includes those receiving 3% Elamipretide in both eyes
Arm/Group | Part A Elamipretide 1.0% Ophthalmic Solution or Placebo | Part B Placebo | Part B Elamipretide 3.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 1 | 3
Participants
  Systemic mild TEAEs | 3 | 1 | 2
  Systemic moderate TEAEs | 2 | 0 | 0
  Systemic severe TEAEs | 2 | 0 | 0

3. Primary Outcome: Change From Baseline in Findings From Slit Lamp Examinations (SLE) Part A
Description: Number of participants who had a change from baseline from normal or abnormal not clinically significant, to abnormal clinically significant (CS) findings for slit lamp examinations (SLE) for Part A. Part B is reported as separate outcome since unit of measure is number of eyes.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, and Week 16
Population: All participants for whom slit lamp outcomes were measured.
Measure: Number; unit: participants
Groups:
- Part A Placebo: Part A Placebo participants received vehicle in paired eye to treatment eye.
- Part A Elamipretide 1.0% Ophthalmic Solution: Part A participants includes those receiving 1% Elamipretide in a randomly selected treatment eye
Arm/Group | Part A Placebo | Part A Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
participants
  Lids Week 1 | 0 | 0
  Lids Week 4: number analyzed (Participants) | 17 | 17
  Lids Week 4 | 0 | 0
  Lids Week 8: number analyzed (Participants) | 17 | 17
  Lids Week 8 | 0 | 0
  Lids Week 12: number analyzed (Participants) | 16 | 16
  Lids Week 12 | 0 | 0
  Lids Week 16: number analyzed (Participants) | 16 | 16
  Lids Week 16 | 0 | 0
  Conjunctiva Week 1 | 0 | 0
  Conjunctiva Week 4: number analyzed (Participants) | 17 | 17
  Conjunctiva Week 4 | 0 | 0
  Conjunctiva Week 8: number analyzed (Participants) | 17 | 17
  Conjunctiva Week 8 | 0 | 0
  Conjunctiva Week 12: number analyzed (Participants) | 16 | 16
  Conjunctiva Week 12 | 0 | 0
  Conjunctiva Week 16: number analyzed (Participants) | 16 | 16
  Conjunctiva Week 16 | 0 | 0
  Cornea Week 1 | 1 | 1
  Cornea Week 4: number analyzed (Participants) | 17 | 17
  Cornea Week 4 | 0 | 0
  Cornea Week 8: number analyzed (Participants) | 17 | 17
  Cornea Week 8 | 1 | 1
  Cornea Week 12: number analyzed (Participants) | 16 | 16
  Cornea Week 12 | 1 | 1
  Cornea Week 16: number analyzed (Participants) | 16 | 16
  Cornea Week 16 | 1 | 1
  Anterior Chamber Week 1 | 0 | 0
  Anterior Chamber Week 4: number analyzed (Participants) | 17 | 17
  Anterior Chamber Week 4 | 0 | 0
  Anterior Chamber Week 8: number analyzed (Participants) | 17 | 17
  Anterior Chamber Week 8 | 0 | 0
  Anterior Chamber Week 12: number analyzed (Participants) | 16 | 16
  Anterior Chamber Week 12 | 0 | 0
  Anterior Chamber Week 16: number analyzed (Participants) | 16 | 16
  Anterior Chamber Week 16 | 0 | 0
  Posterior Chamber Week 1 | 0 | 0
  Posterior Chamber Week 4: number analyzed (Participants) | 17 | 17
  Posterior Chamber Week 4 | 0 | 0
  Posterior Chamber Week 8: number analyzed (Participants) | 17 | 17
  Posterior Chamber Week 8 | 0 | 0
  Posterior Chamber Week 12: number analyzed (Participants) | 16 | 16
  Posterior Chamber Week 12 | 0 | 0
  Posterior Chamber Week 16: number analyzed (Participants) | 16 | 16
  Posterior Chamber Week 16 | 0 | 0
  Iris Week 1 | 0 | 0
  Iris Week 4: number analyzed (Participants) | 17 | 17
  Iris Week 4 | 0 | 0
  Iris Week 8: number analyzed (Participants) | 17 | 17
  Iris Week 8 | 0 | 0
  Iris Week 12: number analyzed (Participants) | 16 | 16
  Iris Week 12 | 0 | 0
  Iris Week 16: number analyzed (Participants) | 16 | 16
  Iris Week 16 | 0 | 0
  Lens Week 1 | 0 | 0
  Lens Week 4: number analyzed (Participants) | 17 | 17
  Lens Week 4 | 0 | 0
  Lens Week 8: number analyzed (Participants) | 17 | 17
  Lens Week 8 | 0 | 0
  Lens Week 12: number analyzed (Participants) | 16 | 16
  Lens Week 12 | 0 | 0
  Lens Week 16: number analyzed (Participants) | 16 | 16
  Lens Week 16 | 0 | 0

4. Primary Outcome: Change From Baseline in Findings From Slit Lamp Examinations (SLE) Part B
Description: Number of eyes with a change from baseline from normal or abnormal not clinically significant, to abnormal clinically significant (CS) findings for slit lamp examinations (SLE) for Part B. Part A is reported as separate outcome.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, and Week 16
Population: All participants for whom slit lamp outcomes were measured with both baseline and post-baseline measurements.
Measure: Number; unit: participants
Units Other Than Participants: eyes
Groups:
- Part B Placebo: Part B Placebo participants received vehicle in both eyes.
Arm/Group | Part B Placebo | Part B Elamipretide 3.0% Ophthalmic Solution
Number analyzed (Participants) | 1 | 3
Number analyzed (eyes) | 2 | 6
participants
  Lids Week 1 | 0 | 0
  Lids Week 4 | 0 | 0
  Lids Week 8: number analyzed (Participants) | 1 | 2
  Lids Week 8: number analyzed (eyes) | 2 | 4
  Lids Week 8 | 0 | 0
  Lids Week 12: number analyzed (Participants) | 1 | 1
  Lids Week 12: number analyzed (eyes) | 2 | 2
  Lids Week 12 | 0 | 0
  Lids Week 16: number analyzed (Participants) | 1 | 1
  Lids Week 16: number analyzed (eyes) | 2 | 2
  Lids Week 16 | 0 | 0
  Conjunctiva Week 1 | 0 | 0
  Conjunctiva Week 4 | 0 | 2
  Conjunctiva Week 8: number analyzed (Participants) | 1 | 2
  Conjunctiva Week 8: number analyzed (eyes) | 2 | 4
  Conjunctiva Week 8 | 0 | 0
  Conjunctiva Week 12: number analyzed (Participants) | 1 | 1
  Conjunctiva Week 12: number analyzed (eyes) | 2 | 2
  Conjunctiva Week 12 | 0 | 0
  Conjunctiva Week 16: number analyzed (Participants) | 1 | 1
  Conjunctiva Week 16: number analyzed (eyes) | 2 | 2
  Conjunctiva Week 16 | 0 | 0
  Cornea Week 1 | 0 | 6
  Cornea Week 4 | 0 | 0
  Cornea Week 8: number analyzed (Participants) | 1 | 2
  Cornea Week 8: number analyzed (eyes) | 2 | 4
  Cornea Week 8 | 0 | 0
  Cornea Week 12: number analyzed (Participants) | 1 | 1
  Cornea Week 12: number analyzed (eyes) | 2 | 2
  Cornea Week 12 | 0 | 0
  Cornea Week 16: number analyzed (Participants) | 1 | 1
  Cornea Week 16: number analyzed (eyes) | 2 | 2
  Cornea Week 16 | 0 | 0
  Anterior Chamber Week 1 | 0 | 0
  Anterior Chamber Week 4 | 0 | 0
  Anterior Chamber Week 8: number analyzed (Participants) | 1 | 2
  Anterior Chamber Week 8: number analyzed (eyes) | 2 | 4
  Anterior Chamber Week 8 | 0 | 0
  Anterior Chamber Week 12: number analyzed (Participants) | 1 | 1
  Anterior Chamber Week 12: number analyzed (eyes) | 2 | 2
  Anterior Chamber Week 12 | 0 | 0
  Anterior Chamber Week 16: number analyzed (Participants) | 1 | 1
  Anterior Chamber Week 16: number analyzed (eyes) | 2 | 2
  Anterior Chamber Week 16 | 0 | 0
  Posterior Chamber Week 1 | 0 | 0
  Posterior Chamber Week 4 | 0 | 0
  Posterior Chamber Week 8: number analyzed (Participants) | 1 | 2
  Posterior Chamber Week 8: number analyzed (eyes) | 2 | 4
  Posterior Chamber Week 8 | 0 | 0
  Posterior Chamber Week 12: number analyzed (Participants) | 1 | 1
  Posterior Chamber Week 12: number analyzed (eyes) | 2 | 2
  Posterior Chamber Week 12 | 0 | 0
  Posterior Chamber Week 16: number analyzed (Participants) | 1 | 1
  Posterior Chamber Week 16: number analyzed (eyes) | 2 | 2
  Posterior Chamber Week 16 | 0 | 0
  Iris Week 1 | 0 | 0
  Iris Week 4 | 0 | 0
  Iris Week 8: number analyzed (Participants) | 1 | 2
  Iris Week 8: number analyzed (eyes) | 2 | 4
  Iris Week 8 | 0 | 0
  Iris Week 12: number analyzed (Participants) | 1 | 1
  Iris Week 12: number analyzed (eyes) | 2 | 2
  Iris Week 12 | 0 | 0
  Iris Week 16: number analyzed (Participants) | 1 | 1
  Iris Week 16: number analyzed (eyes) | 2 | 2
  Iris Week 16 | 0 | 0
  Lens Week 1 | 0 | 0
  Lens Week 4 | 0 | 0
  Lens Week 8: number analyzed (Participants) | 1 | 2
  Lens Week 8: number analyzed (eyes) | 2 | 4
  Lens Week 8 | 0 | 0
  Lens Week 12: number analyzed (Participants) | 1 | 1
  Lens Week 12: number analyzed (eyes) | 2 | 2
  Lens Week 12 | 0 | 0
  Lens Week 16: number analyzed (Participants) | 1 | 1
  Lens Week 16: number analyzed (eyes) | 2 | 2
  Lens Week 16 | 0 | 0

5. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) for Part A
Description: Change from Baseline in intraocular pressure (IOP) using Goldmann applanation tonometry for Part A
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12
Population: All participants for whom intraocular pressure was measured. Part B is reported as a separate Outcome Measure.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- Placebo Part A: Part A: Each subject will receive one drop of vehicle ophthalmic solution BID in the fellow control eye.
  Placebo A: Placebo for Part A
- Elamipretide 1.0% Ophthalmic Solution: Cohort A Each subject will receive one drop of elamipretide 1.0% ophthalmic solution in the randomly selected study eye BID.
  Part A Elamipretide 1.0% Ophthalmic Solution: Each subject will receive one drop of Elamipretide 1.0% ophthalmic solution in the randomly selected study eye BID.
Arm/Group | Placebo Part A | Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
mmHg
  Week 1 | -0.6 (0.64) | -0.4 (0.49)
  Week 4: number analyzed (Participants) | 17 | 17
  Week 4 | -0.3 (0.47) | -0.2 (0.31)
  Week 8: number analyzed (Participants) | 17 | 17
  Week 8 | -1.1 (0.47) | -0.2 (0.64)
  Week 12: number analyzed (Participants) | 16 | 16
  Week 12 | -0.4 (0.45) | -0.4 (0.43)
  Over All 12 Weeks: number analyzed (Participants) | 16 | 16
  Over All 12 Weeks | -0.6 (0.22) | -0.3 (0.21)

6. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) for Part B
Description: Change from Baseline in intraocular pressure (IOP) using Goldmann applanation tonometry for Part B. Part A is reported separately.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12 , and Week 16 or early discontinuation visit
Population: All participants for whom intraocular pressures were measured.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Groups:
- Placebo Part B: Part B: Each subject will receive one drop of vehicle ophthalmic solution BID in both eyes.
- Elamipretide 3.0% Ophthalmic Solution: Part B Elamipretide 3.0% Ophthalmic Solution: Each subject will receive one drop of Elamipretide 3.0% ophthalmic solution in both eyes BID.
Arm/Group | Placebo Part B | Elamipretide 3.0% Ophthalmic Solution
Number analyzed (Participants) | 1 | 3
Number analyzed (Eyes) | 2 | 6
mmHg
  Week 1 | 3.0 (0.00) | 0.2 (3.19)
  Week 4 | 2.0 (0.00) | -0.8 (1.33)
  Week 8: number analyzed (Participants) | 1 | 2
  Week 8: number analyzed (Eyes) | 2 | 4
  Week 8 | 1.5 (2.12) | 0.8 (1.89)
  Week 12: number analyzed (Participants) | 1 | 1
  Week 12: number analyzed (Eyes) | 2 | 2
  Week 12 | 0.0 (0.00) | 3.5 (2.12)
  Week 16: number analyzed (Participants) | 1 | 1
  Week 16: number analyzed (Eyes) | 2 | 2
  Week 16 | 3.5 (2.12) | 1.0 (1.41)

7. Secondary Outcome: Change From Baseline in Central Corneal Thickness by Visit Part A as Measured by Pachymetry for Part A
Description: Change from Baseline in Central Corneal Thickness by Visit as measured by Pachymetry for Part A. Part B is reported as a separate outcome measure.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, and Week 16
Population: All participants for whom central corneal thickness was measured. Part B is reported as a separate Outcome Measure.
Measure: Mean (Standard Deviation); unit: µm
Groups:
- Placebo Eye - Pachymetry: Part A: Each subject will receive one drop of vehicle ophthalmic solution BID in the fellow control eye.
- Elamipretide 1.0% Ophthalmic Solution Eye-Pachymetry; Elamipretide 1.0% Ophthalmic Solution-Pentacam: Part A Elamipretide 1.0% Ophthalmic Solution: Each subject will receive one drop of Elamipretide 1.0% ophthalmic solution in the randomly selected study eye BID.
- Vehicle Eye-Pentacam: Part A: Each subject will receive one drop of vehicle ophthalmic solution BID in the fellow control eye.
  Placebo A: Placebo for Part A
Arm/Group | Placebo Eye - Pachymetry | Elamipretide 1.0% Ophthalmic Solution Eye-Pachymetry | Vehicle Eye-Pentacam | Elamipretide 1.0% Ophthalmic Solution-Pentacam
Number analyzed (Participants) | 18 | 18 | 18 | 18
µm
  Week 1 | 15.4 (47.95) | 7.2 (19.99) | 1.8 (19.72) | 2.0 (25.51)
  Week 4: number analyzed (Participants) | 17 | 17 | 17 | 17
  Week 4 | 9.4 (19.61) | 6.1 (14.32) | 4.7 (21.20) | 4.8 (26.52)
  Week 8: number analyzed (Participants) | 17 | 17 | 17 | 17
  Week 8 | 15.4 (16.04) | 13.1 (22.35) | 6.1 (15.23) | 7.6 (9.61)
  Week 12: number analyzed (Participants) | 16 | 16 | 16 | 16
  Week 12 | 12.3 (30.31) | 2.1 (31.80) | -1.8 (28.25) | 0.0 (25.87)
  Week 16: number analyzed (Participants) | 16 | 16 | 16 | 16
  Week 16 | 13.7 (19.50) | 8.4 (17.09) | 6.3 (21.18) | 8.7 (27.75)

8. Secondary Outcome: Central Corneal Thickness Part B
Description: Central Corneal Thickness: by-subject data as measured by Pachymetry and Pentacam. Part A is reported as a separate outcome measure.
Time Frame: Baseline (Day 1), Week 1, Week 4, Week 8, Week 12, and Week 16, or Early discontinuation visit
Population: All participants for whom Central Corneal Thickness was measured. Part A is reported as a separate Outcome Measure.
Measure: Number; unit: µm
Groups:
- OD-Pachymetry: Right Eye by Pachymetry
- OD Pentacam: Right Eye as measured by pentacam
- OS: Pachymetry: Left Eye as measured by Pachymetry
- OD-Pentacam: Left Eye as measured by Pentacam
Arm/Group | OD-Pachymetry | OD Pentacam | OS: Pachymetry | OD-Pentacam
Number analyzed (Participants) | 4 | 4 | 4 | 4
µm
  Participant 201 (Elamipretide) Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 201 (Elamipretide) Baseline (Day 1) | 626 | 593 | 604 | 591.3
  Participant 201 (Elamipretide) Week 1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 201 (Elamipretide) Week 1 | 619 | 613 | 633 | 602.3
  Participant 201(Elamipretide) Week 4: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 201(Elamipretide) Week 4 | 623 | 599 | 646 | 600.3
  Participant 201 (Elamipretide) Week 8: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 201 (Elamipretide) Week 8 | 608 | 624.3 | 607 | 608.6
  Participant 201 (Elamipretide) Week 12: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 201 (Elamipretide) Week 12 | 617 | 608.6 | 623 | 593.6
  Participant 201 (Elamipretide) Week 16: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 201 (Elamipretide) Week 16 | 604 | 598.6 | 620 | 600.6
  Participant 203 (Elamipretide) Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 203 (Elamipretide) Baseline (Day 1) | 620 | 627 | 635 | 622.6
  Participant 203 (Elamipretide) Week 1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 203 (Elamipretide) Week 1 | 607 | 618.3 | 623 | 617.3
  Participant 203 (Elamipretide) Early discontinuation visit: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 203 (Elamipretide) Early discontinuation visit | 639 | 621 | 630 | 622
  Participant 204 (Vehicle) Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 204 (Vehicle) Baseline (Day 1) | 656 | 618.3 | 624 | 604.6
  Participant 204 (Vehicle) Week 1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 204 (Vehicle) Week 1 | 629 | 616.6 | 623 | 608.3
  Participant 204 (Vehicle) Week 4: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 204 (Vehicle) Week 4 | 645 | 631 | 619 | 626
  Participant 204 (Vehicle) Week 8: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 204 (Vehicle) Week 8 | 640 | 646.3 | 631 | 645
  Participant 204 (Vehicle) Week 12 | 634 | 645.3 | 621 | 637.6
  Participant 204 (Vehicle) Week 16 | 646 | 638.3 | 627 | 630
  Participant 205 (Elamipretide) Baseline (Day 1): number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 205 (Elamipretide) Baseline (Day 1) | 655 | 652.6 | 632 | 632
  Participant 205 (Elamipretide) Week 1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 205 (Elamipretide) Week 1 | 664 | 655.6 | 643 | 626.3
  Participant 205 (Elamipretide) Week 4: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 205 (Elamipretide) Week 4 | 650 | 687.6 | 656.3 | 656.3
  Participant 205 (Elamipretide) Early Discontinuation: number analyzed (Participants) | 1 | 1 | 1 | 1
  Participant 205 (Elamipretide) Early Discontinuation | 663 | 660.6 | 645 | 642

9. Secondary Outcome: Change From Baseline Endothelial Cell Hexagonality in Percentage Over All 12 Weeks for Part A
Description: Change From Baseline in Endothelial Cell Hexagonality in Percentage Over All 12 Weeks for Part A. Specular microscopy is a noninvasive photographic technique that allows visualization and analyzation the corneal endothelium. Using computer-assisted morphometry, specular microscopes analyzes the size, shape and population of the endothelial cells. Histologically, healthy corneal cells initially have a hexagonal shape. As endothelial cells die, neighboring cells enlarge to cover the empty space once occupied by the cell. This, in turn, causes the remaining cells to lose their hexagonal shape. Assessments were performed using the flex center and full auto methods for Part A and data from the flex center method was summarized. The flex center method was used for Part B. The percent of Part B is entered as a separate outcome measure. A decrease from baseline in % cell hexagonality means worse outcome, a increase from baseline means better outcome.
Time Frame: Baseline, Week 1, 4, 8, and 12
Population: All participants had images taken; data was analyzed for those whose images were of sufficient quality.
Measure: Least Squares Mean (Standard Deviation); unit: percentage of hexagonality
Arm/Group | Part A Placebo | Part A Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
percentage of hexagonality
  Central Cornea: number analyzed (Participants) | 2 | 2
  Central Cornea | 1.518 (7.1703) | -3.155 (7.2515)
  Nasal Cornea: number analyzed (Participants) | 5 | 6
  Nasal Cornea | -6.812 (4.3912) | -2.952 (4.0223)
  Temporal Cornea: number analyzed (Participants) | 4 | 3
  Temporal Cornea | 0.738 (5.0322) | -0.764 (5.1291)

10. Secondary Outcome: Corneal Endothelial Cell Hexagonality Part B
Description: Corneal Endothelial Cell Hexagonality in Percentage by-subject data: Part B. Data was only listed in weeks where images were good enough quality to quantify. Specular microscopy is a noninvasive photographic technique that allows visualization and analyzation the corneal endothelium. Using computer-assisted morphometry, specular microscopes analyzes the size, shape and population of the endothelial cells. Histologically, healthy corneal cells initially have a hexagonal shape. As endothelial cells die, neighboring cells enlarge to cover the empty space once occupied by the cell. This, in turn, causes the remaining cells to lose their hexagonal shape. The flex center method was used for Part B. A decrease in percent of cell hexagonality from baseline means worse outcome, an increase from baseline means better outcome.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, and Week 16 or early discontinuation visit
Population: All participants for whom Corneal Endothelial Cell Hexagonality was measured. Part A is reported as a separate Outcome Measure. For images with poor quality or too few cells to register, there was no data available.
Measure: Number; unit: µm
Units Other Than Participants: eyes
Groups:
- Right Eye: Right Eye Cell Hexagonality in Percentage
- Left Eye: Left Eye Cell Hexagonality in Percentage
Arm/Group | Right Eye | Left Eye
Number analyzed (Participants) | 4 | 4
Number analyzed (eyes) | 4 | 4
µm
  Participant 201 (Elamipretide) Central Week 16: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Central Week 16: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Central Week 16 | 27.75 | NA — "Poor Quality Images" or "too few cells to register"
  Participant 201 (Elamipretide) Temporal Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Temporal Baseline (Day 1): number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Temporal Baseline (Day 1) | 39.50 | NA — "Poor Quality Images" or "too few cells to register"
  Participant 204 (Vehicle) Central Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Baseline (Day 1): number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Central Baseline (Day 1) | NA — "Poor Quality Images" or "too few cells to register" | 42.00
  Participant 204 (Vehicle) Central Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 1: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Central Week 1 | NA — "Poor Quality Images" or "too few cells to register" | 31.67
  Participant 204 (Vehicle) Central Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 4: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Central Week 4 | NA — "Poor Quality Images" or "too few cells to register" | 30.00
  Participant 204 (Vehicle) Central Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 8: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Central Week 8 | NA — "Poor Quality Images" or "too few cells to register" | 46.17
  Participant 204 (Vehicle) Central Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 12: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Central Week 12 | NA — "Poor Quality Images" or "too few cells to register" | 33.00
  Participant 204 (Vehicle) Central Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 16: number analyzed (eyes) | 4 | 1
  Participant 204 (Vehicle) Central Week 16 | NA — "Poor Quality Images" or "too few cells to register" | 49.50
  Participant 204 (Vehicle) Nasal Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Baseline (Day 1): number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Nasal Baseline (Day 1) | NA — "Poor Quality Images" or "too few cells to register" | 41.50
  Participant 204 (Vehicle) Nasal Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 1: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 1 | NA — "Poor Quality Images" or "too few cells to register" | 48.34
  Participant 204 (Vehicle) Nasal Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 4: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 4 | NA — "Poor Quality Images" or "too few cells to register" | 41.34
  Participant 204 (Vehicle) Nasal Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 8: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 8 | NA — "Poor Quality Images" or "too few cells to register" | 35.84
  Participant 204 (Vehicle) Nasal Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 12: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 12 | NA — "Poor Quality Images" or "too few cells to register" | 14.50
  Participant 204 (Vehicle) Nasal Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 16: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 16 | NA — "Poor Quality Images" or "too few cells to register" | 35.43
  Participant 204 (Vehicle) Temporal Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Baseline (Day 1): number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Temporal Baseline (Day 1) | NA — "Poor Quality Images" or "too few cells to register" | 54.50
  Participant 204 (Vehicle) Temporal Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 1: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 1 | NA — "Poor Quality Images" or "too few cells to register" | 30.50
  Participant 204 (Vehicle) Temporal Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 8: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 8 | NA — "Poor Quality Images" or "too few cells to register" | 34.00
  Participant 204 (Vehicle) Temporal Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 12: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 12 | NA — "Poor Quality Images" or "too few cells to register" | 50.00
  Participant 204 (Vehicle) Temporal Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 16: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 16 | NA — "Poor Quality Images" or "too few cells to register" | 45.00

11. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Using the Early Treatment Diabetic Retinopathy Study (ETDRS) Scale for Part A.
Description: Best corrected visual acuity (BCVA) using the using the Early Treatment Diabetic Retinopathy Study (ETDRS) scale by visit. ETDRS charts present a series of five letters of equal difficulty on each row, with standardized spacing between letters and rows; there is a total of 14 lines (70 letters), with letter size increasing further geometrically and equivalently in every line by a factor of 1.2589 (or 0.1 log unit), moving up the chart. Minimum score of zero, maximum score of 100. Change from baseline: a more negative score is worse outcome, a more positive score is better outcome. A lower score means less letters were read correctly (worse outcome) and a higher score means more letters were read correctly (better outcome). Part B was listed separately.
Time Frame: Baseline, Weeks 1, 4, 8, 12, and 16
Population: All participants for whom BCVA score was measured.
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Part A Placebo | Part A Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
letters
  Week 1 | 1.8 (3.51) | 2.3 (4.69)
  Week 4: number analyzed (Participants) | 17 | 17
  Week 4 | 0.8 (5.67) | -0.1 (8.96)
  Week 8: number analyzed (Participants) | 17 | 17
  Week 8 | 2.5 (4.87) | 1.3 (8.11)
  Week 12: number analyzed (Participants) | 16 | 16
  Week 12 | 2.6 (4.59) | 0.8 (6.72)
  Week 16: number analyzed (Participants) | 16 | 16
  Week 16 | 3.8 (5.33) | 2.6 (5.94)

12. Secondary Outcome: Best Corrected Visual Acuity (BCVA) Score Using ETDRS Scale for Part B
Description: Best corrected visual acuity (BCVA) using the using the Early Treatment Diabetic Retinopathy Study (ETDRS) scale by visit. ETDRS charts present a series of five letters of equal difficulty on each row, with standardized spacing between letters and rows; there is a total of 14 lines (70 letters), with letter size increasing further geometrically and equivalently in every line by a factor of 1.2589 (or 0.1 log unit), moving up the chart. Minimum score of zero, maximum score of 100. Change from baseline: a more negative score is worse outcome, a more positive score is better outcome. A lower score means less letters were read correctly (worse outcome) and a higher score means more letters were read correctly (better outcome).
Time Frame: Baseline, Weeks 1, 4, 8, 12, and 16
Population: All participants for whom BCVA score was measured.
Measure: Number; unit: letters
Groups:
- Right Eye; Left Eye: Subjects were randomized to receive one drop of elamipretide 3.0% topical ophthalmic solution BID in both the right and left study eyes or one drop of vehicle topical ophthalmic solution BID in both the right and left eyes.
Arm/Group | Right Eye | Left Eye
Number analyzed (Participants) | 4 | 4
letters
  Participant 201 (Elamipretide) Baseline: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Baseline | 66 | 69
  Participant 201 (Elamipretide) Week 1: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 1 | 62 | 68
  Participant 201 (Elamipretide) Week 4: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 4 | 64 | 62
  Participant 201 (Elamipretide) Week 8: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 8 | 67 | 70
  Participant 201 (Elamipretide) Week 12: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 12 | 68 | 73
  Participant 201 (Elamipretide) Week 16: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 16 | 62 | 63
  Participant 203 (Elamipretide) Baseline: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) Baseline | 63 | 59
  Participant 203 (Elamipretide) Week 1: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) Week 1 | 60 | 60
  Participant 203 (Elamipretide) Unscheduled Visit: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) Unscheduled Visit | 0 | 0
  Participant 203 (Elamipretide) Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) Early Discontinuation | 60 | 57
  Participant 204 (Vehicle) Baseline: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Baseline | 79 | 71
  Participant 204 (Vehicle) Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 1 | 78 | 71
  Participant 204 (Vehicle) Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 4 | 79 | 72
  Participant 204 (Vehicle) Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 8 | 76 | 70
  Participant 204 (Vehicle) Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 12 | 80 | 69
  Participant 204 (Vehicle) Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 16 | 81 | 68
  Participant 205 (Elamipretide) Baseline: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Baseline | 68 | 31
  Participant 205 (Elamipretide) Week 1: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Week 1 | 69 | 30
  Participant 205 (Elamipretide) Week 4: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Week 4 | 63 | 36
  Participant 205 (Elamipretide) Unscheduled: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Unscheduled | NA — Not measured | NA — Not measured
  Participant 205 (Elamipretide) Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Early Discontinuation | 70 | 37

13. Secondary Outcome: Change From Baseline in Endothelial Cell Density Over All 12 Weeks for Part A
Description: Change From Baseline in Endothelial Cell Counts, or density (Counts/mm^2) over all 12 weeks for Part A. Part B is entered as a separate outcome measure.
Time Frame: Baseline, Weeks 1, 4, 8, and 12
Population: All participants for whom endothelial cell counts were measured. All participants had images taken; data was analyzed for those whose images were of sufficient quality.
Measure: Least Squares Mean (Standard Error); unit: counts/mm^2
Arm/Group | Part A Placebo | Part A Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
counts/mm^2
  Central Cornea: number analyzed (Participants) | 2 | 2
  Central Cornea | 11.0 (224.89) | -166.9 (231.84)
  Nasal Cornea: number analyzed (Participants) | 5 | 6
  Nasal Cornea | -68.9 (114.22) | -33.0 (105.18)
  Temporal Cornea: number analyzed (Participants) | 4 | 3
  Temporal Cornea | -38.0 (162.07) | -24.0 (178.93)

14. Secondary Outcome: Corneal Endothelial Cell Density Part B
Description: Corneal Endothelial Cell Density: Part B, By-subject data for all time points where images were readable. For all time points where there were "Poor Quality Images" or "too few cells to register", there were no data available, and these were not listed below.
Time Frame: Baseline, Weeks 1, 4, 8, 12, and 16.
Population: All participants for whom Corneal Endothelial Cell Counts/Density was measured. Part A is reported as a separate Outcome Measure. All images from Participant 205 were "poor quality images" and hence, no data was available.
Measure: Number; unit: counts/mm^2
Groups:
- Right Eye: Right Eye Cell Corneal Endothelial Cell Density
- Left Eye: Left Eye Cell Corneal Endothelial Cell Density
Arm/Group | Right Eye | Left Eye
Number analyzed (Participants) | 4 | 4
counts/mm^2
  Participant 201 (Elamipretide) Central Week 16: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Central Week 16 | 934.0 | NA — "Poor Quality Images" or "too few cells to register"
  Participant 201 (Elamipretide) Temporal Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Temporal Baseline (Day 1) | 1449.0 | NA — "Poor Quality Images" or "too few cells to register"
  Participant 204 (Vehicle) Central Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Baseline (Day 1) | NA — Poor Quality Images" or "too few cells to register" | 1241.7
  Participant 204 (Vehicle) Central Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 1 | NA — Poor Quality Images" or "too few cells to register" | 1069.2
  Participant 204 (Vehicle) Central Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 4 | NA — Poor Quality Images" or "too few cells to register" | 1087.7
  Participant 204 (Vehicle) Central Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 8 | NA — Poor Quality Images" or "too few cells to register" | 1149.5
  Participant 204 (Vehicle) Central Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 12 | NA — Poor Quality Images" or "too few cells to register" | 773.2
  Participant 204 (Vehicle) Central Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 16 | NA — Poor Quality Images" or "too few cells to register" | 1094.5
  Participant 204 (Vehicle) Nasal Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Baseline (Day 1) | NA — Poor Quality Images" or "too few cells to register" | 897.3
  Participant 204 (Vehicle) Nasal Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 1 | NA — Poor Quality Images" or "too few cells to register" | 1361.2
  Participant 204 (Vehicle) Nasal Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 4 | NA — Poor Quality Images" or "too few cells to register" | 971.5
  Participant 204 (Vehicle) Nasal Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 8 | NA — Poor Quality Images" or "too few cells to register" | 995.2
  Participant 204 (Vehicle) Nasal Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 12 | NA — Poor Quality Images" or "too few cells to register" | 961.3
  Participant 204 (Vehicle) Nasal Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 16 | NA — Poor Quality Images" or "too few cells to register" | 1046.7
  Participant 204 (Vehicle) Temporal Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Baseline (Day 1) | NA — Poor Quality Images" or "too few cells to register" | 826.0
  Participant 204 (Vehicle) Temporal Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 1 | NA — Poor Quality Images" or "too few cells to register" | 1195.2
  Participant 204 (Vehicle) Temporal Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 8 | NA — Poor Quality Images" or "too few cells to register" | 1068.3
  Participant 204 (Vehicle) Temporal Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 12 | NA — Poor Quality Images" or "too few cells to register" | 1213.3
  Participant 204 (Vehicle) Temporal Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 16 | NA — Poor Quality Images" or "too few cells to register" | 1032.5

15. Secondary Outcome: Change From Baseline in Endothelial Cell Coefficient of Variation Over All 12 Weeks for Part A
Description: Change From Baseline in Endothelial Cell Coefficient of Variation Over All 12 Weeks. Coefficient of variation (CV) is Standard deviation (SD) of cell area divided by the mean cell area of endothelial cell analyzed. CV represents the coefficient, or degree, of variation in the sizes of the endothelial cells (polymegethism). By measuring the variation in size between endothelial cells, the system can measure how much cell loss is occurring. The more variation, the worse the outcome. Part B is is entered as a separate outcome measure.
Time Frame: Baseline, Week 12
Population: All participants had images taken; data was analyzed for those whose images were of sufficient quality.
Measure: Least Squares Mean (Standard Deviation); unit: SD of cell area/Mean cell area, (μm^2)
Arm/Group | Part A Placebo | Part A Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
SD of cell area/Mean cell area, (μm^2)
  Central Cornea: number analyzed (Participants) | 2 | 2
  Central Cornea | -7.644 (7.7617) | -7.941 (8.0334)
  Nasal Cornea: number analyzed (Participants) | 5 | 6
  Nasal Cornea | -3.809 (3.9095) | -4.293 (3.6388)
  Temporal Cornea: number analyzed (Participants) | 4 | 3
  Temporal Cornea | 7.823 (5.0620) | 0.737 (5.0326)

16. Secondary Outcome: Coefficient of Variation (CoV) Part B
Description: Part B, By-subject data for all time points where images were readable. For all time points where there were "Poor Quality Images" or "too few cells to register" there were no data available. CoV represents the coefficient, or degree, of variation in the sizes of the endothelial cells. By measuring the variation in size between endothelial cells, the system can measure how much cell loss is occurring. A CoV less than 40 is normal.
Time Frame: Baseline, Weeks 1, 4, 8,12, and 16
Population: as for outcome 14
Measure: Number; unit: SD of cell area/Mean cell area, (μm^2)
Arm/Group | Right Eye | Left Eye
Number analyzed (Participants) | 4 | 4
SD of cell area/Mean cell area, (μm^2)
  Participant 201 (Elamipretide) Central Week 16: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Central Week 16 | 64.0 | NA — "Poor Quality Images" or "too few cells to register"
  Participant 201 (Elamipretide) Temporal Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Temporal Baseline (Day 1) | 51.0 | NA — "Poor Quality Images" or "too few cells to register"
  Participant 204 (Vehicle) Central Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Baseline (Day 1) | NA — "Poor Quality Images" or "too few cells to register" | 61.0
  Participant 204 (Vehicle) Central Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 1 | NA — "Poor Quality Images" or "too few cells to register" | 69.0
  Participant 204 (Vehicle) Central Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 4 | NA — "Poor Quality Images" or "too few cells to register" | 47.7
  Participant 204 (Vehicle) Central Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 8 | NA — "Poor Quality Images" or "too few cells to register" | 58.7
  Participant 204 (Vehicle) Central Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 12 | NA — "Poor Quality Images" or "too few cells to register" | 60.2
  Participant 204 (Vehicle) Central Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Central Week 16 | NA — "Poor Quality Images" or "too few cells to register" | 56.8
  Participant 204 (Vehicle) Nasal Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Baseline (Day 1) | NA — "Poor Quality Images" or "too few cells to register" | 73.0
  Participant 204 (Vehicle) Nasal Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 1 | NA — "Poor Quality Images" or "too few cells to register" | 58.7
  Participant 204 (Vehicle) Nasal Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 4 | NA — "Poor Quality Images" or "too few cells to register" | 59.5
  Participant 204 (Vehicle) Nasal Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 8 | NA — "Poor Quality Images" or "too few cells to register" | 51.5
  Participant 204 (Vehicle) Nasal Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 12 | NA — "Poor Quality Images" or "too few cells to register" | 65.0
  Participant 204 (Vehicle) Nasal Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Nasal Week 16 | NA — "Poor Quality Images" or "too few cells to register" | 50.0
  Participant 204 (Vehicle) Temporal Baseline (Day 1): number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Baseline (Day 1) | NA — "Poor Quality Images" or "too few cells to register" | 62.3
  Participant 204 (Vehicle) Temporal Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 1 | NA — "Poor Quality Images" or "too few cells to register" | 58.2
  Participant 204 (Vehicle) Temporal Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 8 | NA — "Poor Quality Images" or "too few cells to register" | 63.0
  Participant 204 (Vehicle) Temporal Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 12 | NA — "Poor Quality Images" or "too few cells to register" | 32.3
  Participant 204 (Vehicle) Temporal Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Temporal Week 16 | NA — "Poor Quality Images" or "too few cells to register" | 63.0

17. Secondary Outcome: Change From Baseline in Corneal Area Affected by Microcysts for Part A
Description: Change from Baseline in corneal area affected by microcysts by visit for Part A.
Time Frame: Baseline, Weeks 1, 4, 8, 12, and 16
Population: All participants for whom corneal area affected by microcysts was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Placebo | Part A Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
Participants
  Week 1 Worsened | 0 | 1
  Week 1 No Change | 18 | 17
  Week 1 Improved | 0 | 0
  Week 4 Worsened: number analyzed (Participants) | 17 | 17
  Week 4 Worsened | 0 | 0
  Week 4 No Change: number analyzed (Participants) | 17 | 17
  Week 4 No Change | 17 | 17
  Week 4 Improved: number analyzed (Participants) | 17 | 17
  Week 4 Improved | 0 | 0
  Week 8 Worsened: number analyzed (Participants) | 16 | 17
  Week 8 Worsened | 1 | 1
  Week 8 No Change: number analyzed (Participants) | 16 | 17
  Week 8 No Change | 16 | 16
  Week 8 Improved: number analyzed (Participants) | 16 | 17
  Week 8 Improved | 0 | 0
  Week 12 Worsened: number analyzed (Participants) | 16 | 16
  Week 12 Worsened | 1 | 2
  Week 12 No Change: number analyzed (Participants) | 16 | 16
  Week 12 No Change | 15 | 14
  Week 12 Improved: number analyzed (Participants) | 16 | 16
  Week 12 Improved | 0 | 0
  Week 16 Worsened: number analyzed (Participants) | 16 | 16
  Week 16 Worsened | 0 | 1
  Week 16 No Change: number analyzed (Participants) | 16 | 16
  Week 16 No Change | 16 | 15
  Week 16 Improved: number analyzed (Participants) | 16 | 16
  Week 16 Improved | 0 | 0

18. Secondary Outcome: Corneal Area Affected by Microcysts: Part B
Description: Corneal area affected by microcysts: by-subject data for Part B. No microcysts were present for any timepoints.
Time Frame: Baseline, Weeks 1, 4, 8, 12, and 16, or early discontinuation visit
Population: All participants for whom corneal area affected by microcysts was measured.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Right Eye: Right Eye Locations affected by microcysts
- Left Eye: Left eye locations affected by microcysts
Arm/Group | Right Eye | Left Eye
Number analyzed (Participants) | 4 | 4
Number analyzed (eyes) | 4 | 4
eyes
  Participant 201 (Elamipretide) All visits: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) All visits: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) All visits | 0 | 0
  Participant 203 (Elamipretide) All visits: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) All visits: number analyzed (eyes) | 1 | 1
  Participant 203 (Elamipretide) All visits | 0 | 0
  Participant 204 (Placebo) All visits: number analyzed (Participants) | 1 | 1
  Participant 204 (Placebo) All visits: number analyzed (eyes) | 1 | 1
  Participant 204 (Placebo) All visits | 0 | 0
  Participant 205 (Elamipretide) All visits: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) All visits: number analyzed (eyes) | 1 | 1
  Participant 205 (Elamipretide) All visits | 0 | 0

19. Secondary Outcome: Change From Baseline in Corneal Bullae for Part A.
Description: Count of participants in number, size and location of bullae by treatment. Part B is listed separately.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, Week 16
Population: All participants for whom corneal bullae were measured.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Vehicle: Part A Placebo participants received vehicle in paired eye to treatment eye.
- Elamipretide 1.0% Ophthalmic Solution: Part A participants includes those receiving 1% Elamipretide in eye paired with Placebo eye
Arm/Group | Part A Vehicle | Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
Participants
  Central Inferior 3 Bullae >1mm, 8 Bullae <0.5mm | 0 | 1
  Central Nasal 3 bullae >1mm, 8 bullae <0.5mm | 0 | 1
  Central (Superior) 3 Bullae >1mm, 8 Bullae <0.5mm | 0 | 1
  Central (Temporal) 3 Bullae >1mm, 8 Bullae <0.5mm | 0 | 1

20. Secondary Outcome: Corneal Bullae: Part B
Description: Number, size and location of Corneal bullae: By-subject data: Part B.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, or early discontinuation visit
Population: All participants for whom corneal bullae were measured.
Measure: Number; unit: number of corneal bullae
Units Other Than Participants: eye
Groups:
- Right Eye: Corneal Bullae in Right Eye
- Left Eye: Corneal Bullae in Left Eye
Arm/Group | Right Eye | Left Eye
Number analyzed (Participants) | 4 | 4
Number analyzed (eye) | 4 | 4
number of corneal bullae
  Participant 201 (Elamipretide ) All weeks: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide ) All weeks: number analyzed (eye) | 1 | 1
  Participant 201 (Elamipretide ) All weeks | 0 | 0
  Participant 203 (Elamipretide) All weeks: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) All weeks: number analyzed (eye) | 1 | 1
  Participant 203 (Elamipretide) All weeks | 0 | 0
  Participant 204 (Vehicle) All weeks: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) All weeks: number analyzed (eye) | 1 | 1
  Participant 204 (Vehicle) All weeks | 0 | 0
  Participant 205 (Elamipretide) All weeks: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) All weeks: number analyzed (eye) | 1 | 1
  Participant 205 (Elamipretide) All weeks | 0 | 0

21. Secondary Outcome: Change From Baseline in Severity of Corneal Stromal Folds for Part A
Description: Change from baseline in severity of corneal stromal folds by visit. Descriptive assessment made by Investigator; severity is not assessed using a scale.
Time Frame: Baseline, Weeks 1, 4, 8, 12, and 16
Population: All participants for whom corneal stromal folds was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Placebo | Part A Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
Participants
  Week 1 Worsened | 1 | 1
  Week 1 No Change | 16 | 15
  Week 1 Improved | 1 | 2
  Week 4 Worsened: number analyzed (Participants) | 17 | 17
  Week 4 Worsened | 1 | 0
  Week 4 No Change: number analyzed (Participants) | 17 | 17
  Week 4 No Change | 14 | 14
  Week 4 Improved: number analyzed (Participants) | 17 | 17
  Week 4 Improved | 2 | 3
  Week 8 Worsened: number analyzed (Participants) | 17 | 17
  Week 8 Worsened | 2 | 2
  Week 8 No Change: number analyzed (Participants) | 17 | 17
  Week 8 No Change | 11 | 11
  Week 8 Improved: number analyzed (Participants) | 17 | 17
  Week 8 Improved | 4 | 4
  Week 12 Worsened: number analyzed (Participants) | 16 | 16
  Week 12 Worsened | 2 | 2
  Week 12 No Change: number analyzed (Participants) | 16 | 16
  Week 12 No Change | 10 | 12
  Week 12 Improved: number analyzed (Participants) | 16 | 16
  Week 12 Improved | 4 | 2
  Week 16 Worsened: number analyzed (Participants) | 16 | 16
  Week 16 Worsened | 2 | 2
  Week 16 No Change: number analyzed (Participants) | 16 | 16
  Week 16 No Change | 11 | 12
  Week 16 Improved: number analyzed (Participants) | 16 | 16
  Week 16 Improved | 3 | 2

22. Secondary Outcome: Severity of Corneal Stromal Folds:Part B
Description: Severity of corneal stromal folds by-subject data by visit. Descriptive assessment made by Investigator in the following categories: Not present, trace, mild.
Time Frame: Baseline, Week 1, 4, 8, 12, and 16, or early discontinuation visit
Population: All participants for whom corneal stromal folds was measured.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Right Eye: Right Eye -Severity of Corneal Stromal Folds
- Left Eye: Left Eye-Severity of Corneal Stromal Folds
Arm/Group | Right Eye | Left Eye
Number analyzed (Participants) | 4 | 4
Number analyzed (eyes) | 4 | 4
eyes
  Participant 201 (Elamipretide) Baseline-Mild: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Baseline-Mild: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Baseline-Mild | 1 | 1
  Participant 201 (Elamipretide) Week 1 - Trace: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 1 - Trace: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Week 1 - Trace | 1 | 0
  Participant 201 (Elamipretide) Week 1 -Mild: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 1 -Mild: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Week 1 -Mild | 0 | 1
  Participant 201 (Elamipretide) Week 4 -Trace: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 4 -Trace: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Week 4 -Trace | 1 | 1
  Participant 201 (Elamipretide) Week 8-Mild: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 8-Mild: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Week 8-Mild | 1 | 0
  Participant 201 (Elamipretide) Week 8- no folds: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 8- no folds: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Week 8- no folds | 0 | 1
  Participant 201 (Elamipretide) Week 12-Trace: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 12-Trace: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Week 12-Trace | 1 | 0
  Participant 201 (Elamipretide) Week 12- no folds: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 12- no folds: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Week 12- no folds | 0 | 1
  Participant 201 (Elamipretide) Week 16 -Trace: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 16 -Trace: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Week 16 -Trace | 1 | 0
  Participant 201 (Elamipretide) Week 16 - no folds present: number analyzed (Participants) | 1 | 1
  Participant 201 (Elamipretide) Week 16 - no folds present: number analyzed (eyes) | 1 | 1
  Participant 201 (Elamipretide) Week 16 - no folds present | 0 | 1
  Participant 203 (Elamipretide) Baseline-no folds present: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) Baseline-no folds present: number analyzed (eyes) | 1 | 1
  Participant 203 (Elamipretide) Baseline-no folds present | 1 | 1
  Participant 203 (Elamipretide) Week 1: no folds present: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) Week 1: no folds present: number analyzed (eyes) | 1 | 1
  Participant 203 (Elamipretide) Week 1: no folds present | 1 | 1
  Participant 203 (Elamipretide) Unscheduled visit: no folds present: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) Unscheduled visit: no folds present: number analyzed (eyes) | 1 | 1
  Participant 203 (Elamipretide) Unscheduled visit: no folds present | 1 | 1
  Participant 203 (Elamipretide) Early discontinuation: no folds present: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) Early discontinuation: no folds present: number analyzed (eyes) | 1 | 1
  Participant 203 (Elamipretide) Early discontinuation: no folds present | 1 | 1
  Participant 204 (Vehicle) Baseline- Trace: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Baseline- Trace: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Baseline- Trace | 1 | 1
  Participant 204 (Vehicle) Week 1: no folds present: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 1: no folds present: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Week 1: no folds present | 1 | 1
  Participant 204 (Vehicle) Week 4: no folds present: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 4: no folds present: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Week 4: no folds present | 1 | 1
  Participant 204 (Vehicle) Week 8: no folds present: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 8: no folds present: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Week 8: no folds present | 1 | 1
  Participant 204 (Vehicle) Week 12: no folds present: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 12: no folds present: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Week 12: no folds present | 1 | 1
  Participant 204 (Vehicle) Week 16: no folds present: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) Week 16: no folds present: number analyzed (eyes) | 1 | 1
  Participant 204 (Vehicle) Week 16: no folds present | 1 | 1
  Participant 205 (Elamipretide) Baseline: Mild: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Baseline: Mild: number analyzed (eyes) | 1 | 1
  Participant 205 (Elamipretide) Baseline: Mild | 1 | 1
  Participant 205 (Elamipretide) Week 1: Mild: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Week 1: Mild: number analyzed (eyes) | 1 | 1
  Participant 205 (Elamipretide) Week 1: Mild | 1 | 1
  Participant 205 (Elamipretide) Week 4: no folds present: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Week 4: no folds present: number analyzed (eyes) | 1 | 1
  Participant 205 (Elamipretide) Week 4: no folds present | 1 | 0
  Participant 205 (Elamipretide) Week 4: trace: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Week 4: trace: number analyzed (eyes) | 1 | 1
  Participant 205 (Elamipretide) Week 4: trace | 0 | 1
  Participant 205 (Elamipretide) Unscheduled visit: No folds present: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Unscheduled visit: No folds present: number analyzed (eyes) | 1 | 1
  Participant 205 (Elamipretide) Unscheduled visit: No folds present | 1 | 0
  Participant 205 (Elamipretide) Unscheduled visit: trace: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Unscheduled visit: trace: number analyzed (eyes) | 1 | 1
  Participant 205 (Elamipretide) Unscheduled visit: trace | 0 | 1
  Participant 205 (Elamipretide) Early discontinuation visit: no folds present: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Early discontinuation visit: no folds present: number analyzed (eyes) | 1 | 1
  Participant 205 (Elamipretide) Early discontinuation visit: no folds present | 1 | 0
  Participant 205 (Elamipretide) Early discontinuation: trace: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) Early discontinuation: trace: number analyzed (eyes) | 1 | 1
  Participant 205 (Elamipretide) Early discontinuation: trace | 0 | 1

23. Secondary Outcome: Change From Baseline in Contrast Sensitivity (Log Score) for Part A
Description: Change from Baseline in contrast sensitivity over all 12 weeks log score at 3, 6, 12, 18 cycles per degree (cpd) using Vector Vision's CSV-1000E. Standard tables for the VectorVision's CSV-1000E model were used to convert linear results to the log values. Lower log scores equals lower contrast sensitivity and worse outcome. Higher log scores mean higher contrast sensitivity and better outcome. For 3cpd, range is 0.7-2.08; 6 cpd: 0.91-2.29; 12 cpd: 0.61-1.99; 18cpd: 0.17-1.55, unless no gratings were visible. If no gratings were visible, .3 log was subtracted from the lowest score for 3, 6, and 12cpd. For 18cpd .01 log was used, or essentially 100% contrast.
Time Frame: Baseline, Week 1, 4, 8, 12 weeks
Population: All participants for whom contrast sensitivity was measured
Measure: Least Squares Mean (Standard Deviation); unit: log score
Arm/Group | Placebo Part A | Elamipretide 1.0% Ophthalmic Solution
Number analyzed (Participants) | 18 | 18
log score
  3 cycles per degree | 0.084 (0.0554) | -0.013 (0.0499)
  6 cycles per degree | 0.193 (0.0745) | 0.111 (0.0374)
  12 cycles per degree | 0.050 (0.0787) | 0.013 (0.0503)
  18 cycles per degree | 0.122 (0.0637) | 0.080 (0.0564)

24. Secondary Outcome: Contrast Sensitivity for Part B; By-subject Data
Description: Contrast Sensitivity log score at 3, 6, 12, 18 cycles per degree (cpd) using Vector Vision's CSV-1000E by-subject data, Part B. Part A is listed separately. Standard tables for the VectorVision's CSV-1000E model were used to convert linear results to the log values. Lower log scores equals lower contrast sensitivity and worse outcome. Higher log scores mean higher contrast sensitivity and better outcome. For 3cpd, range is 0.7-2.08; 6 cpd: 0.91-2.29; 12 cpd: 0.61-1.99; 18cpd: 0.17-1.55, unless no gratings were visible. If no gratings were visible, .3 log was subtracted from the lowest score for 3, 6, and 12cpd. For 18cpd .01 log was used, or essentially 100% contrast.
Time Frame: Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, or early discontinuation visit
Population: All participants for whom contrast sensitivity was measured.
Measure: Number; unit: log score
Arm/Group | Right Eye | Left Eye
Number analyzed (Participants) | 4 | 4
log score
  Participant 203 (Elamipretide) 3 cpd Screening: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 3 cpd Screening | 0.70 | 0.70
  Participant 203 (Elamipretide) 3 cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 3 cpd Week 1 | 1.00 | 1.00
  Participant 203 (Elamipretide) 3 cpd Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 3 cpd Early Discontinuation | 0.70 | 0.70
  Participant 203 (Elamipretide) 6 cpd Screening: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 6 cpd Screening | 0.61 | 0.90
  Participant 203 (Elamipretide) 6 cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 6 cpd Week 1 | 0.90 | 1.20
  Participant 203 (Elamipretide) 6 cpd Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 6 cpd Early Discontinuation | 0.61 | 0.61
  Participant 203 (Elamipretide) 12cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 12cpd Baseline | 0.60 | 0.31
  Participant 203 (Elamipretide) 12cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 12cpd Week 1 | 0.31 | 0.60
  Participant 203 (Elamipretide) 12cpd Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 12cpd Early Discontinuation | 0.60 | 0.60
  Participant 203 (Elamipretide) 18cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 18cpd Baseline | 0.01 | 0.18
  Participant 203 (Elamipretide) 18cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 18cpd Week 1 | 0.01 | 0.18
  Participant 203 (Elamipretide) 18 cpd Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 203 (Elamipretide) 18 cpd Early Discontinuation | 0.01 | 0.18
  Participant 204 (Vehicle) 3cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 3cpd Baseline | 1.18 | 1.18
  Participant 204 (Vehicle) 3cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 3cpd Week 1 | 1.63 | 1.00
  Participant 204 (Vehicle) 3cpd Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 3cpd Week 4 | 1.49 | 1.34
  Participant 204 (Vehicle) 3cpd Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 3cpd Week 8 | 1.49 | 1.34
  Participant 204 (Vehicle) 3cpd Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 3cpd Week 12 | 1.79 | 1.63
  Participant 204 (Vehicle) 3cpd Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 3cpd Week 16 | 1.79 | 1.34
  Participant 204 (Vehicle) 6cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 6cpd Baseline | 1.38 | 1.38
  Participant 204 (Vehicle) 6cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 6cpd Week 1 | 1.85 | 1.20
  Participant 204 (Vehicle) 6cpd Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 6cpd Week 4 | 1.38 | 1.56
  Participant 204 (Vehicle) 6cpd Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 6cpd Week 8 | 1.70 | 1.20
  Participant 204 (Vehicle) 6cpd Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 6cpd Week 12 | 1.70 | 1.56
  Participant 204 (Vehicle) 6cpd Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 6cpd Week 16 | 2.00 | 0.90
  Participant 204 (Vehicle) 12cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 12cpd Baseline | 0.60 | 0.60
  Participant 204 (Vehicle) 12cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 12cpd Week 1 | 1.08 | 0.90
  Participant 204 (Vehicle) 12cpd Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 12cpd Week 4 | 1.26 | 1.08
  Participant 204 (Vehicle) 12cpd Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 12cpd Week 8 | 0.60 | 0.90
  Participant 204 (Vehicle) 12cpd Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 12cpd Week 12 | 1.08 | 0.60
  Participant 204 (Vehicle) 12cpd Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 12cpd Week 16 | 1.26 | 0.60
  Participant 204 (Vehicle) 18cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 18cpd Baseline | 0.65 | 0.01
  Participant 204 (Vehicle) 18cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 18cpd Week 1 | 0.65 | 0.18
  Participant 204 (Vehicle) 18cpd Week 4: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 18cpd Week 4 | 0.65 | 0.65
  Participant 204 (Vehicle) 18cpd Week 8: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 18cpd Week 8 | 0.18 | 0.48
  Participant 204 (Vehicle) 18cpd Week 12: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 18cpd Week 12 | 0.65 | 0.01
  Participant 204 (Vehicle) 18cpd Week 16: number analyzed (Participants) | 1 | 1
  Participant 204 (Vehicle) 18cpd Week 16 | 0.65 | 0.65
  Participant 205 (Elamipretide) 3cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 3cpd Baseline | 1.34 | 0.40
  Participant 205 (Elamipretide) 3cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 3cpd Week 1 | 1.18 | 0.40
  Participant 205 (Elamipretide) 3cpd Week 4: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 3cpd Week 4 | 0.70 | 0.40
  Participant 205 (Elamipretide) 3cpd Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 3cpd Early Discontinuation | 1.00 | 0.40
  Participant 205 (Elamipretide) 6cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 6cpd Baseline | 0.90 | 0.61
  Participant 205 (Elamipretide) 6cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 6cpd Week 1 | 0.90 | 0.61
  Participant 205 (Elamipretide) 6cpd Week 4: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 6cpd Week 4 | 0.61 | 0.61
  Participant 205 (Elamipretide) 6cpd Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 6cpd Early Discontinuation | 0.61 | 0.61
  Participant 205 (Elamipretide) 12cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 12cpd Baseline | 0.31 | 0.31
  Participant 205 (Elamipretide) 12cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 12cpd Week 1 | 1.26 | 0.31
  Participant 205 (Elamipretide) 12cpd Week 4: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 12cpd Week 4 | 0.31 | 0.31
  Participant 205 (Elamipretide) 12cpd Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 12cpd Early Discontinuation | 0.31 | 0.31
  Participant 205 (Elamipretide) 18cpd Baseline: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 18cpd Baseline | 0.01 | 0.01
  Participant 205 (Elamipretide) 18cpd Week 1: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 18cpd Week 1 | 0.65 | 0.01
  Participant 205 (Elamipretide) 18cpd Week 4: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 18cpd Week 4 | 0.01 | 0.01
  Participant 205 (Elamipretide) 18cpd Early Discontinuation: number analyzed (Participants) | 1 | 1
  Participant 205 (Elamipretide) 18cpd Early Discontinuation | 0.01 | 0.01

ADVERSE EVENTS:
Time Frame: From the screening period (Day-28 to Day 1) to Week 16 follow up visit, approximately 5 months in total.
Groups:
- Part A Elamipretide 1.0% Ophthalmic Solution and Placebo: Part A participants includes those receiving 1% Elamipretide in one eye and placebo in other eye. This arm will report systemic events that cannot be attributed to either intervention.
- Part A Placebo Only: These will be reporting ocular AEs for placebo eye only. Part A participants includes those receiving Placebo in one eye only.
- Part A Elamipretide 1.0% Ophthalmic Solution Only: These will be reporting ocular AEs for elamipretide eye only. Part A participants includes those receiving 1% Elamipretide in one eye only.
- Part B Placebo: Part B participants includes those receiving Placebo in both eyes. This arm will be reporting ocular and systemic events.
- Part B Elamipretide 3.0% Ophthalmic Solution: Part B participants includes those receiving 3% Elamipretide in both eyes. This arm will be reporting ocular and systemic events.
Arm/Group | Part A Elamipretide 1.0% Ophthalmic Solution and Placebo | Part A Placebo Only | Part A Elamipretide 1.0% Ophthalmic Solution Only | Part B Placebo | Part B Elamipretide 3.0% Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18 | 0/18 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 7/18 | 3/18 | 6/18 | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Elamipretide 1.0% Ophthalmic Solution and Placebo (N=18) | Part A Placebo Only (N=18) | Part A Elamipretide 1.0% Ophthalmic Solution Only (N=18) | Part B Placebo (N=1) | Part B Elamipretide 3.0% Ophthalmic Solution (N=3)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Elamipretide 1.0% Ophthalmic Solution and Placebo (N=18) | Part A Placebo Only (N=18) | Part A Elamipretide 1.0% Ophthalmic Solution Only (N=18) | Part B Placebo (N=1) | Part B Elamipretide 3.0% Ophthalmic Solution (N=3)
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 0
Dry Eye (Eye disorders) | 0 | 1 | 1 | 1 | 0
Conjunctival Haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye pruritis (Eye disorders) | 0 | 0 | 1 | 0 | 1
Eyelid Oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 2
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Eye Pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vital dye staining cornea present (Investigations) | 0 | 2 | 1 | 0 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increase (Investigations) | 1 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Investigations) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Cardioversion (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Shoulder arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Eyelid Disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0
Cataract Cortical (Eye disorders) | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT02653391/Prot_SAP_000.pdf